CLINICAL TRIAL: NCT06702150
Title: Effect of the Primary Nursing Model on Health Outcomes of Elderly Person with Multimorbidity: a Quasi-experimental Study
Brief Title: Nursing Model and Health Outcomes of Elderly People with Multimorbidity: a Quasi-experimental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital da Luz, Portugal (Other)
Collaborators: Universidade Católica Portuguesa (Other)
Responsible Party: Principal Investigator, Isabel Gonçalves, Head of nursing, Hospital da Luz, Portugal
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CES/01/2022/ME
Record Dates: First submitted 2024-11-12; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Multimorbidity; Aged; Patient Outcome Assessment

STUDY DESIGN:
Intervention Model Description: In the hospital where the study was carried out, each nurse is responsible for the whole care of a group of people on one working day and may or may not be given responsibility for the same people on subsequent days (individualized care model). An intervention was proposed in an inpatient unit consisting of implementing the model of organizing care by primary nursing in which a nurse is responsible for the care plan for a group of people from admission to discharge from the unit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Changing the nursing care model to the primary nursing model (Experimental): Inpatient unit where the primary nursing model has been implemented.
  Interventions: Behavioral: Changing the nursing care model to the primary nursing model
- Standard of care (No Intervention): In this unit there was no change in the model of nursing care; the model used was the individualized care model. In this model, each nurse is responsible for the whole care of a group of patients on one working day and may or may not be given responsibility for the same patients on subsequent days. The patients who agreed to participate in the study completed the same questionnaires and at the same frequency as the patients in the intervention unit.

INTERVENTIONS:
Behavioral: Changing the nursing care model to the primary nursing model — The nurses received training in primary nursing care before the start of the intervention. The model was tested and implemented in early April 2022. Since then, all patients admitted to the unit have been assigned to a primary nurse within the first 48 hours. This nurse is responsible for developing and monitoring the patient's care plan, assessing care needs, implementing the care plan and evaluating the outcomes. This nurse is also responsible for coordinating care needs and discharge planning with other healthcare professionals. When the primary nurse is not working, another nurse from his or her team continues the care plan that he or she has defined. All patients admitted to the unit who met the selection criteria were informed about the study and, if they agreed to take part, completed a self-care competence questionnaire at admission (baseline), at discharge and one month after discharge. They also completed a questionnaire on satisfaction with nursing care at discharge.
  Arms: Changing the nursing care model to the primary nursing model

SUMMARY:
The goal of this quasi-experimental study is to analyze the effect of organizing nursing care according to the primary nursing model on therapeutic self-care and satisfaction with nursing care for elderly people with multimorbidity in hospital. Participants were patients of both sexes aged over 65 years with at least two chronic diseases admitted to an acute hospital ward. The main questions it aims to answer are:

* Does the use of the primary nursing model increase participants' perceived ability for therapeutic self-care?
* Does the use of the primary care model increase participants' satisfaction with nursing care? The researchers are comparing whether implementing the primary nursing model with the usual care model increases patients' capacity for therapeutic self-care.

Participants:

* Complete a self-care skills questionnaire on admission to the inpatient unit;
* Complete the same self-care questionnaire on discharge from hospital;
* Complete the same self-care questionnaire by telephone one month after discharge from hospital
* Complete a nursing care satisfaction questionnaire on discharge from hospital;

DETAILED DESCRIPTION:
The self-care skills questionnaire used was the Therapeutic Self-care Scale (TSC), translated and validated for the Portuguese population.

The questionnaire used to assess satisfaction with care was the Scale of Citizen Satisfaction with Care (ESCCE), validated for the Portuguese population.

ELIGIBILITY:
Inclusion Criteria:

* Have at least two chronic diseases
* Have at least one disease classified in the International Classification of Diseases, Ninth Revision (ICD9) and belonging to one of the following groups: cardiovascular disease, cancer, chronic obstructive pulmonary disease and diabetes;
* Expect to be hospitalised for more than 48 hours;
* Have the cognitive ability to read, write and understand the information provided;
* Speak, read and write Portuguese.

Exclusion Criteria:

* Transfer to other levels of care within the organisation
* Discharged to other care units outside the organisation
* Episodes of readmission within 30 days of leaving hospital, as this made the last moment of data collection impossible.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 206 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Average global self-care score at discharge from inpatient unit | On the day of discharge from the inpatient unit, assessment up to 24 hours later.
  Evaluated by the difference in response to the Therapeutic Self-Care Scale on admission and discharge from the unit. It is a 12-question Likert scale with a minimum score of zero (0) and a maximum score of five (5), with higher scores corresponding to better results. Average response scores are used.
Average global self-care score at follow-up | At the follow-up 30 days after hospital discharge
  Evaluated by the difference between the response to the Therapeutic Self-Care Scale at discharge and at follow-up.
  Also assessed by the difference between the response to the Therapeutic Self-Care Scale at admission and at follow-up.
  Therapeutic Self-Care Scale is a 12-question Likert scale with a minimum score of zero (0) and a maximum score of five (5), with higher scores corresponding to better results. Average response scores are used.

SECONDARY OUTCOMES:
Average score for satisfaction with nursing care at discharge from inpatient unit | On the day of discharge from the inpatient unit, assessment up to 24 hours later.
  Assessed by answering the Citizen Satisfaction with Nursing Care Scale at discharge from the unit. This is a 47-question Likert scale with a minimum score of one (1) and a maximum of seven (7), with higher scores corresponding to better results. Average and total response scores are used.

CONTACTS AND LOCATIONS:
Overall Officials: Elvio Jesus, Professor, Study Director — Universidade Católica Portuguesa; Elisabete Nunes, Professor, Study Chair — Nursing School of Lisbon
Locations (1):
- Hospital da LUz, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: SAP

REFERENCES:
- [Derived] Goncalves I, Almeida S, Jesus E, Nunes E. Effect of the Primary Nursing Model on Self-Care Skills of Hospitalized Older Patients with Multimorbidity: A Quasi-Experimental Study. Healthcare (Basel). 2025 Sep 27;13(19):2457. doi: 10.3390/healthcare13192457. PMID 41095543